CLINICAL TRIAL: NCT06173518
Title: A Single-Arm, Open-Label, Multi-Centre, Phase Ib Study Evaluating the Safety and Preliminary Efficacy of AUTO1 in Pediatric Patients With CD19-Positive Relapsed/ Refractory (r/r) B Cell Acute Lymphoblastic Leukemia (B ALL) and Aggressive Mature B Cell Non-Hodgkin Lymphoma (B NHL)
Brief Title: A Study of CD19 Targeted CAR T Cell Therapy in Pediatric Patients With Relapsed or Refractory B Cell Acute Lymphoblastic Leukemia (B ALL) and Aggressive Mature B-cell Non-Hodgkin Lymphoma (B NHL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO1-PY1; 2023-506307-26-00 (Other: EU CT)
Record Dates: First submitted 2023-12-08; First posted 2023-12-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Relapsed or Refractory B Cell Acute Lymphoblastic Leukemia; Relapsed or Refractory B Cell Non-Hodgkin Lymphoma
Keywords: B cell acute lymphoblastic leukemia; B cell Non-Hodgkin lymphoma; Relapsed B cell acute lymphoblastic leukemia; Relapsed B cell Non-Hodgkin lymphoma; Refractory B cell acute lymphoblastic leukemia; Refractory B cell Non-Hodgkin lymphoma; Aggressive mature B cell Non-Hodgkin lymphoma; Pediatric ALL; Pediatric NHL; AUTO1; Obecabtagene autoleucel; CD19-positive CAR T cell; Obe-cel
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma; Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUTO1 (Experimental)
  Interventions: Biological: AUTO1

INTERVENTIONS:
Biological: AUTO1 — Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with anti-CD19 chimeric antigen receptor (CAR) T cells
  Other Names: Obecabtagene autoleucel (obe-cel)

SUMMARY:
This is a Phase Ib study to evaluate the safety and efficacy of autologous T cells engineered with a chimeric antigen receptor (CAR) targeting cluster of differentiation (CD)19 in pediatric patients with relapsed or refractory (r/r) B cell acute lymphoblastic leukemia (B ALL) and r/r B cell Non-Hodgkin lymphoma (B NHL)

DETAILED DESCRIPTION:
This is a single-arm, open-label, multi-center, Phase Ib study to determine the safety and preliminary efficacy of obe-cel administered intravenously in pediatric patients with r/r B ALL and with r/r aggressive mature B NHL. This study is designed to evaluate the safety and preliminary efficacy of obe-cel.

The safety and tolerability of obe-cel in pediatric patients will be continually monitored by the Sponsor. Additionally, the Independent Data Monitoring Committee (IDMC) will review the rolling safety data generated after 6 and 12 treated patients have been monitored for at least 28 days and every 6 months thereafter, and in the event any protocol defined safety stopping criteria are met. If no pre-defined safety events related to obe-cel are met, and the safety data are consistent with what has previously been observed with obe-cel, the IDMC can recommend continuing the study without or with modifications. Based on emerging data, the study may be stopped early due to excessive toxicity, i.e., certain pre-defined obe-cel-related safety events or deaths.

The study will involve consented patients going through the following sequential study periods: screening, leukapheresis, bridging as necessary, lymphodepletion, treatment evaluation, and follow-up.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female patients < 18 years old at screening
* Patients with ≥ 6 kg body weight at screening

B ALL Cohort: r/r CD19-positive B ALL defined as:

1. Primary refractory disease defined as:

   1. National Cancer Institute high risk (defined as presenting with white blood cell count ≥ 50 × 10^9 cells/L or aged ≥ 10 years at diagnosis) patients with MRD ≥ 0.01% after first-line induction and consolidation and blinatumomab (if allowed per country specific approvals and treatment guidelines).
   2. Refractory B ALL if BM disease ≥ 25% after first line induction and consolidation.
   3. KMT2A rearranged infant ALL with MRD ≥ 1% after first line induction and blinatumomab (if allowed per country specific approvals and treatment guidelines) or MRD ≥ 0.01% after first line induction and consolidation.
2. First relapse

   1. Children's Oncology Group high risk first relapse involving BM < 36 months after initial diagnosis or an isolated extramedullary relapse < 18 months after initial diagnosis.
   2. Patients with Down syndrome and infants with KMT2A rearranged are eligible with first relapse at any time.
   3. Refractory disease with MRD ≥ 0.01% after re-induction for first relapse (with or without blinatumomab, if allowed per country specific approvals and treatment guidelines).
3. Second or greater relapse
4. Relapsed or refractory post-SCT:

   a. Relapsed or refractory disease after allogeneic transplant provided obe cel infusion occurs ≥ 3 months after SCT.
5. Philadelphia chromosome positive (Ph+) ALL:

   1. Any of the above with Ph+ ALL where patient is intolerant to or has failed at least one tyrosine kinase inhibitor (TKI) or if TKI therapy is contraindicated.

B NHL Cohort: r/r CD19-positive aggressive mature B NHL defined as 1 of the following:

1. Relapsed after one or more prior therapies (can include allogeneic and autologous hematopoietic SCT).
2. Primary refractory (have not achieved a CR or PR after the first line of therapy) with measurable, disease by radiological criteria at screening including the B NHL subtypes: (i) diffuse large B-cell lymphoma (DLBCL), (ii) Burkitt's lymphoma, (iii) primary mediastinal large B-cell lymphoma (PMBCL) and (iv) high-grade B-cell lymphoma (not otherwise specified).

   * Karnofsky (age ≥ 10 years) or Lansky (age < 10 year) performance status score ≥ 50%.
   * In patients with B ALL, local documentation of CD19 expression on leukemic blasts in the BM, peripheral blood, or cerebrospinal fluid (CSF) or biopsy done no more than 30 days prior to consent. In patients treated with blinatumomab, testing should be undertaken after blinatumomab therapy has been stopped. In patients with mature B NHL, CD19 expression must be confirmed in a biopsy after any CD19 targeted therapies.
   * Adequate renal, hepatic, pulmonary, and cardiac function.

EXCLUSION CRITERIA:

* Diagnosis of chronic myelogenous leukemia lymphoid in blast crisis.
* History or presence of clinically relevant central nervous system (CNS) pathology unrelated to CNS leukemia.
* Presence of CNS-3 disease or CNS-2 disease with neurological changes at screening.
* Presence of active or uncontrolled fungal, bacterial, viral, or other infection requiring systemic antimicrobials for management.
* Patients who had prior (< 3 months before obe-cel infusion) stem cell transplant.
* Prior CD19 targeted therapy other than blinatumomab.
* Patients who have experienced Grade ≥ 3 neurotoxicity following blinatumomab.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
Incidence and duration of severe hypogammaglobulinemia | Up to 24 months

SECONDARY OUTCOMES:
Overall remission rate (ORR) in B ALL patients | Up to 24 months
  Defined as best response of complete remission (CR) or complete remission with incomplete recovery of counts (CRi) per Investigator assessment occurring at any time after obe-cel infusion
Overall response rate (ORR) in B NHL patients | Up to 24 months
  Defined as best response of complete response (CR) or partial response (PR) per Investigator assessment occurring at any time after obe-cel infusion
Duration of remission (DOR) in B ALL | Up to 24 months
Duration of response (DOR) in B NHL | Up to 24 months
Overall survival (OS) in B ALL | Up to 24 months
Overall survival (OS) in B NHL | Up to 24 months
Incidence of CD19-negative relapse at any time in B ALL | Up to 24 months
Incidence of CD19-negative relapse at any time in B NHL | Up to 24 months
Event-free survival (EFS) in B ALL | Up to 24 months
Proportion of patients achieving minimal residual disease (MRD)-negative remission in bone marrow (BM) within 3 months of obe-cel dosing in B ALL | Up to 24 months
Proportion of patients achieving complete remission (CR) within 3 months per Investigator assessment in B ALL | Up to 24 months
Progression-free survival (PFS) in B NHL | Up to 24 months
Proportion of patients undergoing stem cell transplantation (SCT) while still in CR/CRi following obe-cel (in B ALL) | Up to 24 months
Proportion of enrolled patients for whom an obe-cel product can be manufactured and administered. | Up to 6 months post-leukapheresis
Detection of CAR T cells (copies/μg genomic deoxyribonucleic acid) measured by droplet digital polymerase chain reaction in the peripheral blood and BM following obe-cel infusion including duration of detectability. | Up to 24 months
Quantification of depletion of circulating CD19 expressing B cells as determined by flow cytometry in the peripheral blood. | Up to 24 months
Frequency and duration of hospitalization and/or critical care support to manage obe-cel-related toxicity within 6 months of obe-cel dosing. | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Methodist Children's Hospital, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Nino Jesus, Madrid
- United Kingdom (3):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester
  - Great North Children's Hospital, Newcastle upon Tyne